CLINICAL TRIAL: NCT06451068
Title: Assistive Robotically Aligning Optical Coherence Tomography of the Retinal Periphery
Brief Title: Peripheral Retina Robotically Aligned OCT Study
Acronym: PR-RAOCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00115348; R21EY033959 (NIH)
Record Dates: First submitted 2024-06-05; First posted 2024-06-10 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Retinal Disease
Keywords: Optical Coherence Tomography (OCT)
MeSH Terms: conditions — Retinal Diseases | interventions — Tomography, Optical Coherence; Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to a group based on ocular history/diagnosis. Each participant will receive the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Group 1 - Healthy adult volunteers (Experimental): Healthy adult volunteers recruited from the patient population, students or employees of Duke University or Duke Eye Center (n=7)
  Interventions: Device: Peripheral retina robotically aligned optical coherence tomography (OCT) system; Other: Likert Scales
- Group 2 - Adult participants with "flashers and floaters" (Experimental): Adult participants recruited from the patient population of Duke Eye Center with complaints of "flashers and floaters" undergoing clinical examination (n=7)
  Interventions: Device: Peripheral retina robotically aligned optical coherence tomography (OCT) system; Other: Likert Scales
- Group 3 - Adult participants with flashers and floaters with no diagnosed peripheral retinal breaks (Experimental): Adult participants recruited from the patient population of Duke Eye Center with complaints of "flashers and floaters" and a clinical examination showing no breaks in the peripheral retina (n=22)
  Interventions: Device: Peripheral retina robotically aligned optical coherence tomography (OCT) system; Other: Likert Scales
- Group 4 - Adult participants with flashers and floaters with diagnosed peripheral retinal breaks (Experimental): Adult participants recruited from the patient population of Duke Eye Center with complaints of "flashers and floaters" and a clinical examination showing one or more breaks in the peripheral retinal (n=22)
  Interventions: Device: Peripheral retina robotically aligned optical coherence tomography (OCT) system; Other: Likert Scales

INTERVENTIONS:
Device: Peripheral retina robotically aligned optical coherence tomography (OCT) system — To visualize the full 360° of the retinal periphery (from equator to the more anterior ora serrata), investigators developed and redesigned a conical mirror contact lens and our non-contact robotically aligning platform to deliver OCT to the peripheral retina. The peripheral retina robotically aligned OCT (PR-RAOCT) system is built around a 6-axis cooperative robot (UR5e, Universal Robots), using our previously developed RAOCT control software.
  Other Names: PR-RAOCT
Other: Likert Scales — Survey evaluating relative comfort with each type of peripheral exam (scleral depression vs. PR-RAOCT). Participants will rate 3 items on a 1 (non) to 5 (maximum) Likert scale: overall discomfort, physical pain, and photophobia for each exam.

SUMMARY:
Optical coherence tomography (OCT) is a 3D imaging technology that has seen wide adoption within ophthalmology. However, optical access to the retinal periphery remains a challenge for conventional OCT systems. The study team plans to innovate peripheral retinal OCT imaging technology by first developing the first robotic OCT system capable of autonomously assisting the operator during imaging of the human peripheral retina using 3D active tracking and compensation and then by developing of the first OCT system designed for treatment of the retinal periphery.

DETAILED DESCRIPTION:
Purpose and Objectives:

The long-term goal is to develop a system that provides 360° visualization of the peripheral retina replacing the current standard of care for evaluation of the retinal periphery for breaks: indirect ophthalmoscopy with scleral depression, a procedure requiring the examiner to mechanically indent the eye at multiple locations and use an indirect ophthalmoscope and condensing lens to attempt to visualize the retina peripherally and over360°. The rationale for this project is that in addition to being extremely uncomfortable for the patient, this technique requires considerable skill with specialized training.

Furthermore, the exam does not create a direct record of the findings - the examiner must illustrate a guide map from memory for subsequent laser photocoagulation (LP) therapy utilizing this same manual technique. These objectives will be achieved by pursuing two specific aims: 1) Adapt a custom conical mirror contact lens and robotically aligning platform to optically access the peripheral retina with OCT and laser photocoagulation therapy; and 2) Validate peripheral retina robotically aligning OCT against scleral depressed exam in eyes with and without peripheral retinal breaks requiring treatment.

To validate our imaging technique, the investigators will conduct a powered study in eyes with and without known peripheral retina breaks comparing total number of detected peripheral retinal breaks per eye by Peripheral Retina Robotically Aligned OCT (PR-RAOCT) versus clinical exam. As a secondary outcome, the investigators will evaluate subject comfort level following each method. The investigators will recruit patients presenting at the Duke Eye Center with complaints of "flashers and floaters" and have undergone indirect ophthalmoscopy with scleral depression as part of their standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able and willing to consent to study participation
* Subject is more than 18 years of age
* Healthy adult volunteers without known ocular issues other than refractive error

Exclusion Criteria:

* Subject is unwilling or unable to provide consent
* Subject is less than 18 years of age
* Students or employees under direct supervision of the investigators
* Subjects with eye trauma, infection of the anterior ocular tissues or corneal conditions like keratoconus, Peter's anomaly, corneal edema, dense cataracts obscuring the retina and dense capsule opacities in pseudophakes

The investigators will not exclude subjects based on eyes being phakic, pseudo-phakic, or aphakic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Presence of peripheral retinal break/s - Optical Coherence Tomography (OCT) | Single imaging session (day 1)
  Presence of peripheral retinal break as measured by OCT reading
Presence of peripheral retinal break/s - clinical exam | Single imaging session (day 1)
  Presence of peripheral retinal break as measured by clinical exam

SECONDARY OUTCOMES:
Location of peripheral break | Single imaging session (day 1)
  Peripheral break quadrant location (superior, inferior, temporal, nasal) for each exam as seen on OCT.
Comfort evaluation | Single session (day 1)
  Participants will complete a survey evaluating relative comfort with each type of peripheral exam. Participants will rate three items on a 1(none) to 5(maximum) Likert scale. Lower Likert scores equate to a negative response (less comfortable) and a higher Likert score equates to a more positive response (more comfortable).

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Toth, MD, Principal Investigator — Duke University Eye Center
Locations (1):
- Duke University Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No